CLINICAL TRIAL: NCT02930863
Title: Prevention of Post Operative Hypoxia in the Post Anesthesia Care Unit Using Pulse Oximetry With Automated Verbal Prompts
Brief Title: Pulse Oximetry With Automated Verbal Prompts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201600061
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Non-Automated Group (Active Comparator): Participants assigned to this group will receive the standard of care procedures for the monitoring and treatment of hypoxemia. Complete brief post-PACU stay survey.
  Interventions: Behavioral: Brief post-PACU stay survey.
- Automated Prompt Group (Experimental): Participants assigned to this group will utilize the automated verbal prompts to enable their ability to improve their current condition by following generated commands. Complete a questionnaire focused around their experience with the pulse oximetry software and its effects on the patient's satisfaction and experience.
  Interventions: Other: pulse oximetry software; Behavioral: Brief post-PACU stay survey.

INTERVENTIONS:
Other: pulse oximetry software — This pulse oximetry software will utilize automated verbal prompts that direct the patients to breathe when their pulse oximetry reading falls at or below 93%.
  Arms: Automated Prompt Group
Behavioral: Brief post-PACU stay survey. — Complete a brief post-PACU stay survey focused around their satisfaction and experience during their time in the PACU.

SUMMARY:
This study will evaluate the effectiveness of an automated voice prompting system on post operative hypoxia within the Postoperative Anesthesia Care Unit (PACU). This will be done to detect an improvement of the patient experience and provider care through a decrease in the number of peripheral capillary oxygen saturation (SpO2) monitor alarms via the patients own ability to follow the instruction and improve their SpO2 levels.

DETAILED DESCRIPTION:
The investigators will examine and observe the patient's stay in the PACU and utilize the pulse oximetry software and data to analyze the ability to evaluate the difference in patient oxygenation levels and supplemental oxygen use with automated verbal prompted monitoring versus a standard care control group. As well as determine if automated verbal prompted monitoring leads to less monitor alarms and subsequent improvement of subjective alarm fatigue and patient satisfaction with their care versus standard care.

The pulse oximeter will have a finger probe that will be attached to the patient's middle finger to read the patient's SpO2 levels. Each time the participant's pulse oximetry value declines to 93% or less, an automated verbal prompt, created via the software, will generate as a soft prompt. This will be followed up by a hard prompt if no improvement is seen in their oxygenation level after a period of time. A positive feedback elicitation will be given if the participant's saturation levels increase above 93%. This automated verbal prompt guidance will take place during the entirety of the investigational group's PACU stay.

ELIGIBILITY:
Inclusion Criteria:

* planned general anesthetic
* ability to provide informed consent

Exclusion Criteria:

* use of regional anesthesia
* altered mental status
* hearing impairment requiring assistive devices
* inability to hear normal conversational voice during the consent process
* inability preoperatively to squeeze probe finger against thumb for any reason
* baseline SpO2 less than or equal to 93% (on room air or baseline home oxygen requirement)
* history of methemoglobinemia
* suspected or confirmed carbon monoxide (CO) poisoning
* planned admission to an intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of a participant's SpO2 level falling below 87% | Change from baseline up to 24 hours
  SpO2 will be monitored using the standard pulse oximeter system

SECONDARY OUTCOMES:
Change between the study groups number of pulse oximetry alarms | Change from baseline up to 24 hours
  SpO2 will be monitored using the standard physiologic monitoring system
Change between the study groups level of alarm fatigue | Change from baseline up to 24 hours
  Number of participants reporting a decreased level of alarm noise
Change between the study groups level of postoperative care satisfaction | Change from baseline up to 24 hours
  Number of participants reporting alarm noise affected their level of postoperative care satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Samsun Lampotang, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No